CLINICAL TRIAL: NCT05188742
Title: Sequencing and Combination of Mirabegron and Transcutaneous Tibial Nerve Stimulation (TTNS) in Overactive Bladder Syndrome: a Multicenter, Randomized, Open-label, Crossover Trial
Brief Title: Sequencing and Combination of Mirabegron and TTNS in Overactive Bladder Syndrome: a Multicenter, Randomized, Open-label, Crossover Trial
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2021-09-003B
Record Dates: First submitted 2021-11-22; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Overactive Bladder Syndrome
Keywords: overactive bladder; mirabegron; transcutaneous tibial nerve stimulation
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — mirabegron

STUDY DESIGN:
Intervention Model Description: Treatment sequence: randomized with 1:1 ratio to either Sequence A or Sequence B Sequence A: mirabegron 50mg monotherapy x 8 weeks -> multi-modal combination treatment x 4 weeks -> TTNS monotherapy x 8 weeks Sequence B: TTNS monotherapy x 8 weeks -> multi-modal combination treatment x 4 weeks -> mirabegron 50mg monotherapy x 8 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence A (Experimental): mirabegron 50mg OD x 8 weeks, followed by mirabegron 50mg OD and TTNS for 4 weeks, followed by TTNS twice a week x 8 weeks
  Interventions: Drug: mirabegron; Procedure: TTNS
- Sequence B (Experimental): TTNS twice a week x 8 weeks, followed by mirabegron 50mg OD and TTNS for 4 weeks, followed by mirabegron 50mg OD x 8 weeks
  Interventions: Drug: mirabegron; Procedure: TTNS

INTERVENTIONS:
Drug: mirabegron — mirabegron 50mg QD
Procedure: TTNS — transcutaneous tibial nerve stimulation

SUMMARY:
Research question:

A wealth of existing research has established the independent effectiveness of mirabegron and neuromodulation in the treatment of overactive bladder syndrome. Optimizing the use of these effective and well-tolerated treatment modalities is an important clinical goal and warrants further research. The primary aim of this trial is to answer the questions: how does varying the treatment sequence involving mirabegron and transcutaneous tibial nerve stimulation (TTNS) affect efficacy and patient acceptance and what is the second-line efficacy of either treatment modality?

Primary objective:

To evaluate improvement in storage symptoms, as measured by changes in Overactive Bladder Symptom Score (OABSS), International Prostate Symptom Score (IPSS) and parameters of voiding diary, in overactive bladder (OAB) patients receiving mirabegron or TTNS as first-line therapy when crossed over to second-line therapy with the opposite treatment modality

Secondary objectives:

To evaluate improvement in symptoms, as measured by changes in OABSS, IPSS and parameters of voiding diary, on first-line therapy with mirabegron or TTNS followed by combination multi-modal therapy To evaluate the effect of multi-modal treatment approach on patient's perception of treatment satisfaction and symptom control To evaluate urodynamic profiles of patients treated with multi-modal approach

DETAILED DESCRIPTION:
Study design: Prospective, randomized, multicenter, open-label, cross-over trial Treatment sequence: randomized with 1:1 ratio to either Sequence A or Sequence B

Sequence A: mirabegron 50mg monotherapy x 8 weeks -> multi-modal combination treatment x 4 weeks -> TTNS monotherapy x 8 weeks Sequence B: TTNS monotherapy x 8 weeks -> multi-modal combination treatment x 4 weeks -> mirabegron 50mg monotherapy x 8 weeks

Patient population: adults ≥ 20 years who have experienced symptoms of OAB, as defined by International Continence Society (ICS) diagnostic criteria, for at least 3 months

Sample size: approximately 180 patients

ELIGIBILITY:
Inclusion Criteria:

* Adult OAB patients ≥20 years
* Diagnosed with moderate to severe OAB (with or without urgency incontinence) based on OABSS >5 and clinical assessment, with UUI-predominant presentation, for at least 3 months
* Able to receive TTNS and accommodate treatment logistics (30 min per on-site session, twice weekly)
* Provided informed consent to participate in the study

Exclusion Criteria:

* Neurologic conditions associated with OAB symptoms
* History of stress urinary incontinence
* Use of intravesical onabotulinumoxinA within recent 6 months
* Postvoid residual urine volume (PVR) ≥ 100mL
* Evidence of active urinary tract infection or urinary tract stone at screening
* Genitourinary tract operation during the 3-month period prior to baseline
* Confirmed or suspected genitourinary tract or pelvic malignancy
* History of uncontrolled hypertension (systolic >160 mmHg and/or diastolic >110 mmHg)
* History of intolerance to mirabegron
* Patients with pacemakers or implantable defibrillators
* Patients prone to excessive bleeding
* Patients with nerve damage that could impact percutaneous tibial nerve or pelvic floor function
* Patients who are pregnant or planning to become pregnant during the duration of treatment
* History of medical conditions or presence of patient factors that, in the judgement of the investigator, would preclude adherence to study protocol

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-11-10 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline to end of treatment (EoT) (Week 20) in OABSS | Baseline and Week 20
  Changes from baseline to Week 20 in OABSS (Overactive Bladder Symptom Score) (a lower OABSS score represents a better outcome). Symptom improvement is defined as OABSS total score decreased by ≥ 3 points at EoT

SECONDARY OUTCOMES:
Changes from baseline to Week 12 in OABSS | Baseline and Week 12
  Changes from baseline to Week 12 in OABSS (Overactive Bladder Symptom Score) (a lower OABSS score represents a better outcome)
Changes from baseline to Week 12 and 20/end of treatment (EoT) in IPSS | Baseline, and Week 12 and 20
  Changes from baseline in IPSS (International Prostate Symptom Score) at Week 12 and 20 (a lower IPSS represents a better outcome)
Change from Baseline to Week 12 and 20/end of treatment (EoT) in Mean Number of Micturitions per 24 Hours | Baseline, and Week 12 and 20
  The average number of micturitions (urinations) per 24 hours is derived from the number of times a patient urinates (excluding incontinence only episodes) per day recorded by the patient in a micturition diary for 3-days prior to clinic visits at Baseline and Week 12 and 20/end of treatment (EoT).
Change from Baseline to Week 12 and 20/end of treatment (EoT) in Mean Number of Nocturia Episodes per 24 Hours | Baseline, and Week 12 and 20
  Nocturia is defined as waking at night one or more times to void. The average number of times a patient urinates (excluding incontinence only episodes) during sleeping time per day is derived from a micturition diary in which a patient records for 3 days prior to clinic visits at Baseline and Week 12 and 20/end of treatment (EoT).
Change from Baseline to Week 12 and 20/end of treatment (EoT) in Mean Number of Urgency Episodes per 24 Hours | Baseline, and Week 12 and 20
  The average number of urgency episodes (the sudden, compelling desire to pass urine that is difficult to defer) is derived from episodes reocrded by the patient in a micturition diary in which a patient completes for 3 days prior to clinic visits at Baseline and Week 12 and 20/end of treatment (EoT).
Change from Baseline to Week 12 and 20/end of treatment (EoT) in Mean Number of Urgency Incontinence Episodes per 24 Hours | Baseline, and Week 12 and 20
  The involuntary leakage of urine accompanied or immediately proceeded by urgency, derived from the number of incontinence episodes recorded by the patient in a micturition diary in which a patient completes for 3 days prior to clinic visits at Baseline and Week 12 and 20/end of treatment (EoT).
Changes from Week 8 to Week 20 in OABSS | Week 8 to Week 20
  Changes from Week 8 to Week 20 in OABSS (Overactive Bladder Symptom Score) (a lower OABSS represents a better outcome)
Changes from Week 8 to Week 20 in IPSS | Week 8 to Week 20
  Changes from Week 8 to Week 20 in IPSS (International Prostate Symptom Score) (a lower IPSS represents a better outcome)
Changes from Week 8 to Week 20 in Mean Number of Micturitions per 24 Hours | Week 8 to Week 20
  The average number of micturitions (urinations) per 24 hours is derived from the number of times a patient urinates (excluding incontinence only episodes) per day recorded by the patient in a 3-day micturition diary.
Changes from Week 8 to Week 20 in Mean Number of Nocturia Episodes per 24 Hours | Week 8 to Week 20
  Nocturia is defined as waking at night one or more times to void. The average number of times a patient urinates (excluding incontinence only episodes) during sleeping time per day is derived from the 3-day patient micturition diary.
Changes from Week 8 to Week 20 in Mean Number of Urgency Episodes per 24 Hours | Week 8 to Week 20
  The average number of urgency episodes (the sudden, compelling desire to pass urine that is difficult to defer) derived from episodes recorded by the patient in a 3-day micturition diary
Changes from Week 8 to Week 20 in Mean Number of Urgency Incontinence Episodes per 24 Hours | Week 8 to Week 20
  The involuntary leakage of urine accompanied or immediately proceeded by urgency, derived from the number of incontinence episodes recorded by the patient in a 3-day micturition diary
Changes from Week 12 to Week 20 in OABSS | Week 12 to Week 20
  Changes from Week 12 to Week 20 in OABSS (Overactive Bladder Symptom Score) (a lower OABSS represents a better outcome)
Changes from Week 12 to Week 20 in IPSS | Week 12 to Week 20
  Changes from Week 12 to Week 20 in IPSS (International Prostate Symptom Score) (a lower IPSS represents a better outcome)
Changes from Week 12 to Week 20 in Mean Number of Micturitions per 24 Hours | Week 12 to Week 20
  The average number of micturitions (urinations) per 24 hours is derived from the number of times a patient urinates (excluding incontinence only episodes) per day recorded by the patient in a 3-day micturition diary.
Changes from Week 12 to Week 20 in Mean Number of Nocturia Episodes per 24 Hours | Week 12 to Week 20
  Nocturia is defined as waking at night one or more times to void. The average number of times a patient urinates (excluding incontinence only episodes) during sleeping time per day is derived from the 3-day patient micturition diary.
Changes from Week 12 to Week 20 in Mean Number of Urgency Episodes per 24 Hours | Week 12 to Week 20
  The average number of urgency episodes (the sudden, compelling desire to pass urine that is difficult to defer) derived from episodes recorded by the patient in a 3-day micturition diary
Changes from Week 12 to Week 20 in Mean Number of Urgency Incontinence Episodes per 24 Hours | Week 12 to Week 20
  The involuntary leakage of urine accompanied or immediately proceeded by urgency, derived from the number of incontinence episodes recorded by the patient in a 3-day micturition diary
Changes from baseline to Week 12 and 20/end of treatment (EoT) in Overactive Bladder Questionnaire-Short Form (OAB-Q-SF) score | Baseline, and Week 12 and 20
  Overactive Bladder Questionnaire-Short Form (OAB-Q-SF) is a participant-reported instrument consisting of 19 items that assess the degree to which a participant is bothered by OAB symptoms, and the degree of impact of OAB symptoms on daily life. Participants rate each item using a 6-point Likert Scale ranging from "Not at all" to "A very great deal" for the symptom bother items and "none of the time" to "All of the time" for the Health Related Quality of Life (HRQL) items.
Changes from baseline to Week 12 and 20/end of treatment (EoT) in Bladder Assessment Tool (BAT) score | Baseline, and Week 12 and 20
  Bladder Assessment Tool (BAT) is a participant-reported instrument consisting of 17 questions regarding the symptoms, bothering, impacts and treatment satisfaction in the past 7 days. Scores range from 0 to 88, a reduction in BAT score indicates an improvement.
Changes from baseline to Week 12 and 20/end of treatment (EoT) in Treatment Satisfaction-Visual Analog Scale (TS-VAS) score | Baseline, and Week 12 and 20
  Treatment Satisfaction-Visual Analog Scale (TS-VAS) is a quantitative instrument assessing participant improvement in participants with OAB. A score of 10 on the TS-VAS indicates complete satisfaction, whereas a positive change from baseline indicates improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chieh Lin, MD/Phd, Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taipei, Taiwan